CLINICAL TRIAL: NCT05096650
Title: Chang Gung Memorial Hospital, Taipei, Taiwan
Brief Title: Platelet Rich Plasma for Treatment of Facial Photoaging: A Double-blind, Randomized, Split-face Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CMRPG5K0121
Record Dates: First submitted 2021-10-01; First posted 2021-10-27 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-09

CONDITIONS: Platelet-Rich Plasma; Aging
Keywords: Platelet-Rich Plasma; photoaging; mesotherapy

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, split-face
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: 1. The participants will blinded to receive platelet rich plasma and platelet poor plasma injections for treatment of photoaging of right side or left side of face.
  2. The practitioner will inject these blood products into photoaging areas in bilateral face in each case without the knowledge of the content of injection materials.
  3. The outcomes assessors will evaluate the response of the therapies without the knowledge of which blood products injected into bilateral face.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- platelet rich plasma (Experimental): Each case will receive 3 sessions of injection therapies with one month interval. The practitioner will inject 2ml of platelet rich plasma with fan and linear method into photoaging areas in one side of the midface in one session of treatment.
  Interventions: Procedure: mesotherapy of platelet rich plasma and platelet poor plasma
- platelet poor plasma (Other): Each case will receive 3 sessions of injection therapies with one month interval. The practitioner will inject 2ml of platelet rich plasma with fan and linear method into photoaging areas in the other side of the midface in one session of treatment.
  Interventions: Procedure: mesotherapy of platelet rich plasma and platelet poor plasma

INTERVENTIONS:
Procedure: mesotherapy of platelet rich plasma and platelet poor plasma — Each case will receive 3 sessions of injection therapies with one month interval. Each case will receive platelet rich plasma therapy on one side of the face. The other side of the face was treated with platelet poor plasma.

SUMMARY:
Photoaging is characterized by cellular changes and alterations in dermal extracellular matrix proteins with degeneration of connective tissue caused by intrinsic and extrinsic factors. The clinical manifestations of photoaging included wrinkles, pigmented changes, tissue loss, and sagging. Autologous platelet-rich plasma is a preparation of platelets in concentrated plasma from peripheral blood. The α granules of platelets contained many growth factors. According to previous literature, growth factors in platelet-rich plasma directly stimulate fibroblast proliferation to boost collagen production. It has also been shown to modulate extracellular matrix metabolism and remodeling by increasing the expression of specific matrix metalloproteinases. In review of previous literatures, there was only limited researches of platelet-rich plasma for treatment of photoaging. Therefore, the present study was conducted for analyzing the efficacy and safety of autologous platelet-rich plasma in photoaging therapy.

DETAILED DESCRIPTION:
Autologous platelet-rich plasma is a preparation of platelets in concentrated plasma from peripheral blood. The α granules of platelets contained many growth factors, such as platelet-derived growth factor, transforming growth factor, vascular endothelial growth factor, and epithelial growth factor. These growth factors can trigger intracellular signaling cascades that ultimately alter gene expression and protein synthesis. Clinically, autologous platelet-rich plasma has been applied for treatment of hair loss, chronic wounds, and atrophic scars.

Photoaging is characterized by cellular changes and alterations in dermal extracellular matrix proteins with degeneration of connective tissue caused by intrinsic and extrinsic factors. The clinical manifestations of photoaging included wrinkles, pigmented changes, tissue loss, and sagging. The therapeutic modalities of photoaging included energy-based device, filler injection, and surgical treatment. However, there are some limitations and drawbacks of these therapies. For example, filler injection may cause foreign body granuloma, vascular occlusions, or tissue necrosis. Surgical treatment is an invasive procedure which may cause hematoma, infection, or scar formation.

According to previous literature, growth factors in platelet-rich plasma directly stimulate fibroblast proliferation to boost collagen production. It has also been shown to modulate extracellular matrix metabolism and remodeling by increasing the expression of specific matrix metalloproteinases. Platelet-rich plasma-enhanced expression of matrix metalloproteinases -1 and -3 helps clear photodamaged extracellular matrix components and allow for a better quality, more organized collagen meshwork. This process helps soften fine lines and minimize scarring. In addition, transforming growth factor and epithelial growth factor in platelet-rich plasma are known to modulate keratinocyte propagation and migration as well as repair barrier function. In review of previous literatures, there was only limited researches of platelet-rich plasma for treatment of photoaging. Therefore, the present study was conducted for analyzing the efficacy and safety of autologous platelet-rich plasma in photoaging therapy.

ELIGIBILITY:
Inclusion criteria:

1. Men or female patients older than 20 years old with facial photoaging (Glogau Scale type II)
2. The photoaging severity of bilateral face is symmetric.

Exclusion criteria:

1. Patients with thrombocytopenia, coagulopathy, hematopoietic malignancy.
2. Patients with severe inflammation over treated area, malignancy, keloid, or poor wound healing history.
3. Patients had received laser, radiofrequency, ultherapy over treated area within 6 months.
4. Patients had received botulism or filler injection over treated area within 12 months.
5. Patients had received plastic surgery over treated area within 12 months.
6. Patients had severe psychiatric disorders with poor control.
7. Patients with other diseases which are not suitable for receiving platelet rich plasma (PRP) injection therapy.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-11-30 (Estimated); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Global Aesthetic Improvement Scale | 3 months after the last session of treatment
  To assess the global aesthetic improvement in appearance compared to pretreatment (minimum: -1, worse; maximum: 3, very much improved)
Fitzpatrick wrinkle scale | 3 months after the last session of treatment
  To assess the severity of wrinkles of photoaging areas (minimum: 1, mild; maximum: 9, severe)
Wrinkle Severity Rating scale | 3 months after the last session of treatment
  To assess the severity of wrinkles of photoaging areas (minimum: 1, absent; maximum: 5, extreme)

SECONDARY OUTCOMES:
The scores of rhytids in VISIA system | before the 1st, 2nd and 3rd sessions of treatment as well as 1 and 3 months after the last session of treatment
  Apply the scores of different aging domains in VISIA system for evaluating the therapeutic response.
  (minimum: 1, worse; maximum: 100, severe)
The scores of texture in VISIA system | before the 1st, 2nd and 3rd sessions of treatment as well as 1 and 3 months after the last session of treatment
  Apply the scores of different aging domains in VISIA system for evaluating the therapeutic response.
  (minimum: 1, worse; maximum: 100, severe)
The scores of pores size in VISIA system | before the 1st, 2nd and 3rd sessions of treatment as well as 1 and 3 months after the last session of treatment
  Apply the scores of different aging domains in VISIA system for evaluating the therapeutic response.
  (minimum: 1, worse; maximum: 100, severe)
The scores of pigment spots in VISIA system | before the 1st, 2nd and 3rd sessions of treatment as well as 1 and 3 months after the last session of treatment
  Apply the scores of different aging domains in VISIA system for evaluating the therapeutic response.
  (minimum: 1, worse; maximum: 100, severe)
The scores of brownish spots in VISIA system | before the 1st, 2nd and 3rd sessions of treatment as well as 1 and 3 months after the last session of treatment
  Apply the scores of different aging domains in VISIA system for evaluating the therapeutic response.
  (minimum: 1, worse; maximum: 100, severe)

CONTACTS AND LOCATIONS:
Overall Officials: Yau-Li Huang, MD, Principal Investigator — Chang Gung Memorial Hospital, Taipei, Taiwan
Locations (1):
- Chang Gung Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
We will not share IPD due to the privacy of participants.

REFERENCES:
- [Result] Lee ZH, Sinno S, Poudrier G, Motosko CC, Chiodo M, Saia W, Gothard D, Thomson JE, Hazen A. Platelet rich plasma for photodamaged skin: A pilot study. J Cosmet Dermatol. 2019 Feb;18(1):77-83. doi: 10.1111/jocd.12676. Epub 2018 May 31. PMID 29855132
- [Result] Cameli N, Mariano M, Cordone I, Abril E, Masi S, Foddai ML. Autologous Pure Platelet-Rich Plasma Dermal Injections for Facial Skin Rejuvenation: Clinical, Instrumental, and Flow Cytometry Assessment. Dermatol Surg. 2017 Jun;43(6):826-835. doi: 10.1097/DSS.0000000000001083. PMID 28375975
- [Result] Elnehrawy NY, Ibrahim ZA, Eltoukhy AM, Nagy HM. Assessment of the efficacy and safety of single platelet-rich plasma injection on different types and grades of facial wrinkles. J Cosmet Dermatol. 2017 Mar;16(1):103-111. doi: 10.1111/jocd.12258. Epub 2016 Jul 29. PMID 27474688
- [Result] Mehryan P, Zartab H, Rajabi A, Pazhoohi N, Firooz A. Assessment of efficacy of platelet-rich plasma (PRP) on infraorbital dark circles and crow's feet wrinkles. J Cosmet Dermatol. 2014 Mar;13(1):72-8. doi: 10.1111/jocd.12072. PMID 24641609